CLINICAL TRIAL: NCT06731270
Title: Phase II Study of Diclofenac Salvage in Patients Metastatic Non-Small Cell Lung Cancer With Early Signs of Progression on Single Agent PD(L)-1 Blockade
Brief Title: Diclofenac for the Treatment of Patients With Metastatic Non-small Cell Lung Cancer on Single Agent Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Carlisle, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006572; NCI-2024-07760 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00006572 (Other: Emory University Hospital/Winship Cancer Institute); Winship6018-23 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Specimen Handling; cemiplimab; Diclofenac; Magnetic Resonance Spectroscopy; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (diclofenac, immunotherapy) (Experimental): Patients receive diclofenac PO BID and standard of care immunotherapy with pembrolizumab, atezolizumab, nivolumab or cemiplimab on day 1 of each cycle. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and CT, PET, or MRI on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Drug: Diclofenac Potassium; Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Atezolizumab — Given atezolizumab
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given cemiplimab
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Diclofenac Potassium — Given PO
  Other Names: Cambia; Cataflam; CGP 45840B; Zipsor
Other: Electronic Health Record Review — Ancillary studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given nivolumab
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Biological: Pembrolizumab — Given pembrolizumab
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests how well diclofenac works in treating patients non-small cell lung cancer (NSCLC) that may have spread from where it first started (primary site) to other places in the body (metastatic) on single agent immunotherapy. Diclofenac, a type of non-steroidal anti-inflammatory (NSAID), blocks the body's production of a substance that causes inflammation and may decrease tumor growth and improve the effectiveness of immunotherapy. Immunotherapy with pembrolizumab, atezolizumab, nivolumab or cemiplimab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving diclofenac may kill more tumor cells in patients with metastatic NSCLC on single agent immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical benefit rate of concomitant diclofenac potassium (diclofenac) and single agent checkpoint blockade.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of concomitant diclofenac and single agent checkpoint blockade.

II. To evaluate the efficacy of concomitant diclofenac and single agent checkpoint blockade in NSCLC.

EXPLORATORY OBJECTIVES:

I. To evaluate the change in immunophenotype in circulating CD8 T cells following initiation of diclofenac oral therapy in patients who show early sings of progression on single agent immunotherapy for advanced lung cancer.

II. To investigate the role of PD-L1 expression status in response to the addition of diclofenac daily oral therapy in patients who show early sings of progression on single agent immunotherapy for advanced lung cancer.

III. To evaluate the role of serum lactic acid levels in determining dose exposure to diclofenac.

IV. To evaluate the change in circulating immune parameters (CD4 T cells and B cells) with the addition of diclofenac to single agent immunotherapy.

V. To evaluate the role of the tumor microenvironment at the time of diagnosis on efficacy.

OUTLINE:

Patients receive diclofenac orally (PO) twice daily (BID) and standard of care immunotherapy with pembrolizumab, atezolizumab, nivolumab or cemiplimab on day 1 of each cycle. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and computed tomography (CT), positron emission tomography (PET), or magnetic resonance imaging (MRI) on study.

After completion of study treatment, patients are followed up every 12 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Capable of signing informed consent
* Age ≥ 18 years at time of study entry
* Stage III or IV pathologically proven NSCLC with advanced or metastatic disease, currently on treatment with an Food and Drug Administration (FDA) approved single agent monoclonal antibody inhibiting the PD(L)-1 pathway (pembrolizumab, atezolizumab, nivolumab, or cemiplimab) for a minimum of 12 weeks

  * May include frontline single agent immune checkpoint inhibitors (ICI), maintenance single agent ICI after chemo-ICI, or subsequent line therapy
* Radiographic evidence of clinical progression as determined by the treating physician, not warranting immediate change of therapy. Progressive disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria is not required. This can include mixed response, will need at least one growing lesion. Exposure to PD1 inhibitor for at least 12 weeks will minimize the risk of pseudo-progression
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of ≥ 26 weeks
* Absolute neutrophil count (ANC) ≥ 1,000 cell/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8 gm/dL
* Creatinine clearance ≥ 45 ml/ml
* Bilirubin ≤ 1.5 x institutional upper limit of normal

  * Bilirubin must be ≤ 3 x institutional upper limit of normal in patients with documented Gilbert's syndrome
* Serum glutamic oxaloacetic transaminase (SGOT) / serum gluatmic pyruvic transaminase (SGPT) ≤ 2.5 x institutional upper limit of normal
* Ability to take oral medications
* Willingness and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is non-therapeutic
* Prophylactic or therapeutic anticoagulation therapy including but not limited to: warfarin, heparin, low molecular weight heparin, or direct oral anticoagulants, including: dabigatran (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis), edoxaban (Savaysa), and betrixaban (Bevyxxa)
* Treatment within the previous 6 weeks or planned initiation of bevacizumab
* Abnormal markers of coagulation as measured by international normalized ratio (INR) > 2
* Contraindication for NSAID therapy including: chronic aspirin therapy for coronary artery disease (CAD), cerebrovascular accident (CVA), or other indication, uncontrolled gastrointestinal ulcerative disease, known bleeding diathesis, known allergy or hypersensitivity to NSAIDS, advanced renal disease, uncontrolled hypertension, known seizure disorder or others
* Female of childbearing potential unwilling or unable to use 2 methods of contraception, detailed in protocol
* Uncontrolled intercurrent illness
* History of another primary malignancy with exceptions noted in protocol
* History of active primary immunodeficiency or active infection including tuberculosis, hepatitis B, hepatitis C
* Current or prior use of immunosuppressive medication within 14 days before the first dose of diclofenac. There are exceptions to this criterion
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study medications
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | At 12 weeks
  CBR will be defined as complete response, partial response, and/or stable disease. Clinical response will be assessed using Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 criteria. Clinical benefit rate will be reported as a proportion, with an exact 80% confidence interval estimated using the Clopper-Pearson method.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs severity will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Descriptive statistics will be reported, using frequencies and percentages for each toxicity.
Objective response rate (ORR) | At 12 weeks
  ORR will be defined per RECIST 1.1. ORR will be reported as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method.
Progression-free survival (PFS) | From initiation of treatment to progression or death up to 1 year
  PFS will be determined by RECIST 1.1. PFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median PFS will be estimated using the Brookmeyer-Crowley approach.
Overall survival (OS) | From diagnosis to death from any cause up to 1 year
  OS will be estimated using the Kaplan-Meier method, and median OS will be calculated. A 95% confidence interval will be estimated using the Brookmeyer-Crowley approach.
Duration of response (DOR) | From the date of first response to the date of the first progressive disease or death due to any cause up to 1 year
  DOR will be estimated using the Kaplan-Meier method, and median DOR will be calculated. A 95% confidence interval will be estimated using the Brookmeyer-Crowley approach.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W Carlisle, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia